CLINICAL TRIAL: NCT02232555
Title: A Ten-week, Randomized, Double-blind Study Evaluating the Efficacy of Duloxetine 60 mg Once Daily Versus Placebo in Outpatients With Major Depressive Disorder and Pain (EU-Pain Enriched Study)
Brief Title: Study to Evaluate the Efficacy of Duloxetine in Outpatients With Major Depressive Disorder and Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1208.10
Record Dates: First submitted 2014-09-04; First posted 2014-09-05 (Estimated); Last update posted 2014-09-05 (Estimated); Status verified 2014-08

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Duloxetine Hydrochloride

ARMS (2):
- Duloxetine (Experimental)
  Interventions: Drug: Duloxetine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Duloxetine
  Arms: Duloxetine
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study was to investigate the efficacy of duloxetine versus placebo on pain in outpatients with major depressive disorder (MDD): change in Brief Pain Inventory Short Form (BPI-SF) 24-hour average pain score from baseline over the 8 weeks of treatment

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients who meet the criteria for MDD according to the Diagnostic and Statistic Manual of mental disorders, 4th edition (DSM-IV) criteria and confirmed by Mini International Neuropsychiatric Interview (MINI)
* Montgomery-Asberg Depression Rating Scale (MADRS) score ≥20 at screening and baseline (Visits 1 and 2)
* Patients must have had at least one previous episode of depression in their medical history
* Painful physical symptoms (PPS) with a score ≥ 3 on the BPI-SF scale for average pain at screening and baseline
* Patient aged 18 years or older at the screening visit
* CGI-Severity score ≥ 4 at Visits 1 and 2
* Patients willing and able to comply with the scheduled visits, tests and procedures required by the protocol
* Written informed consent obtained at the screening visit, in accordance with Good clinical practice (GCP) and local regulatory requirements, prior to any study procedure

Exclusion Criteria:

Neuro-psychiatric exclusions

* Lack of response of the current episode to 2 or more adequate courses of antidepressant therapy given at a clinically appropriate dose and for a sufficient length of time in the judgement of the investigator
* Any anxiety disorder as a primary diagnosis within the past 6 months (including panic disorder, obsessive-compulsive disorder, posttraumatic stress disorder, generalized anxiety disorder, and social phobia). Note: Specific phobias (i.e. agoraphobia, arachnophobia, etc.) will be allowed
* Any diagnosis of bipolar disorder, schizophrenia, or other psychotic disorders
* Presence of an Axis II disorder which, in the judgement of the investigator, would interfere with compliance with the study protocol
* History of serious suicide attempt or patient judged to be at serious suicidal risk in the opinion of the investigator and / or score > 2 for question 10 (suicide) of the MADRS
* History of drug dependence, including alcohol or benzodiazepines, according to DSM-IV, in the previous year
* Positive urine screen for drug abuse (cannabis, benzodiazepines, barbiturates, opiates, cocaine, amphetamines)

Other medical exclusions

* Patients requiring continuous treatment with analgesics (> step 2 WHO definition) because of chronic pain (> 6 months)
* Patients with organic pain syndromes
* Epilepsy or history of seizure disorder or of a treatment with anticonvulsant medication for epilepsy or seizures
* Patients with a known diagnosis of raised intraocular pressure or at risk of acute narrow-angle glaucoma
* Known diagnosis of congenital galactosaemia, glucose or galactose malabsorption syndrome, or lactose deficiency
* Patients with severely impaired renal function, defined by a creatinine clearance < 30 mL/min (creatinine clearance was calculated by the central laboratory from the screening safety laboratory test
* Acute liver injury (such as hepatitis) or severe (Child-Pugh Class C) cirrhosis
* Abnormal initial ECG findings according to investigator's judgement
* Serious medical illness or clinically significant laboratory abnormalities which, in the judgement of the investigator, are likely to require medication/ intervention or hospitalization during the course of the study
* Women of childbearing potential not using a medically accepted means of contraception when engaging in sexual intercourse (e.g. intrauterine device, oral contraceptive, contraceptive patch, implant, or barrier devices)
* Women who are pregnant or breast-feeding

Pharmacological and other exclusions

* Participation in another clinical trial within 30 days prior to screening (Visit 1)
* Patients who have previously completed or withdrawn from this or any other study investigating duloxetine or have previously been treated with duloxetine
* Treatment with a monoamine oxidase inhibitor (MAOI) within 14 days prior to Visit 2 or potential need to use a MAOI within 5 days after discontinuation of study drug
* Treatment with fluoxetine within 28 days prior to Visit 2
* Treatment with any of excluded medications (listed in Protocol) within 7 days prior to Visit 2

  * (excepted MAOI within 14 days and fluoxetine within 28 days)
* Frequent and/or severe allergic reactions with multiple medications. Known hypersensitivity to duloxetine or any of the inactive ingredients
* Electro-convulsive Therapy (ECT) or Transcranial Magnetic Stimulation (TMS) within one year prior to screening
* Initiation or discontinuation of depression-oriented psychotherapeutic treatment (e.g. behavioural therapy, psychoanalytic therapy, cognitive therapy etc.) within 6 weeks prior to screening visit or planned use of such treatment at any time during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 327
Dates: Start 2005-05; Primary Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Change of 24-hour average pain rated on Brief Pain Inventory-Short Form (BPI-SF) score | Up to 8 weeks after drug administration

SECONDARY OUTCOMES:
Change in Montgomery-Asberg Depression Rating Scale (MADRS) total score | Up to 8 weeks after drug administration
Time to sustained clinical response for Painful Physical Symptoms (PPS) according BPI-SF score | Up to 8 weeks after drug administration
  as defined by 30% reduction from baseline in question 5 (average pain) of the BPI-SF score
Change of patient symptoms rated on Symptom Checklist 90 Revised (SCL-90-R) scale | Up to 8 weeks after drug administration
Patients Global Impression (PGI) rated on PGI-improvement scale | Up to 8 weeks after drug administration
Clinical Global Impressions (CGIs) by investigator rated on CGI-severity score | Up to 8 weeks after drug administration
Clinical Global Impressions (CGIs) by investigator rated on CGI-improvement scale | Up to 8 weeks after drug administration
Time to sustained clinical response for overall depression symptoms | Up to 8 weeks after drug administration
  as defined by a 50% reduction from baseline in MADRS score
Number of patients with adverse events | Up to 8 weeks after drug administration
Number of patients withdrawing due to adverse event | Up to 8 weeks after drug administration
Number of patients with clinical significant findings in vital signs | Up to 8 weeks after drug administration
  blood pressure, pulse rate
Number of patients with clinical significant findings in weight | Up to 8 weeks after drug administration
Number of patients with clinical significant findings in laboratory values | Up to 8 weeks after drug administration